CLINICAL TRIAL: NCT04103788
Title: Evaluation of Increased Absorption of a Curcumin Emulsion (CurQ+) in Healthy Volunteers Either Following Enzymatic Hydrolysis Pre-Treatment or Direct Analysis of Split Serum Samples
Brief Title: Evaluation of Increased Absorption of a Curcumin Emulsion (CurQ+) in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ESM-CLN#2018T01
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Bioavailability
Keywords: Bioavailability; Absorption

STUDY DESIGN:
Intervention Model Description: open-label, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 95% Curcuminoid Powder (Active Comparator): Curcumin powder standardized to >95% curcuminoids, single dose, used to determine standard absorptivity of unformulated powder.
  Interventions: Dietary Supplement: 95% Curcuminoid Powder
- CurQ+ (Experimental): Highly absorbed curcumin coconut oil emulsion, single dose, used to produce serum samples for analytical comparison of sample preparation methodologies.
  Interventions: Dietary Supplement: CurQ+

INTERVENTIONS:
Dietary Supplement: 95% Curcuminoid Powder — 1200 mg curcuminoids
  Arms: 95% Curcuminoid Powder
Dietary Supplement: CurQ+ — 400 mg curcuminoids + coconut oil + polysorbate
  Arms: CurQ+

SUMMARY:
This study is intended to evaluate the comparative effects of direct analysis of serum samples versus pre-treatment with enzymatic hydrolysis in split samples obtained from dosing with a highly absorbed curcumin emulsion product that is commercially available as BIOCURC.

DETAILED DESCRIPTION:
When curcumin is absorbed by the body, it is primarily found in the bloodstream as curcumin glucuronide (C-gluc) and curcumin sulfate (C-SO4) metabolites. Traditionally bioavailability studies have performed an enzymatic hydrolysis pre-treatment of serum samples with both a glucuronidase and a sulfatase enzyme in order to produce free curcumin for analysis via HPLC. In subsequent years, standards have become available for the metabolites (C-gluc & C-SO4) that make it possible to determine these compound levels directly in serum samples using HPLC-MS-MS. Initial pilot work had indicated that enzymatic hydrolysis was producing falsely elevated results for bioavailability. We wanted to evaluate this in a more formal setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects must be 21-75 years of age at the time of screening.

   a. Female subjects must agree to use one of the following medically acceptable contraceptive methods from the Screening visit (unless otherwise stated) through the End of Study (EOS) visit. Acceptable methods include: abstinence, same-sex partner, double barrier (condom, diaphragm, or cervical cap with spermicidal foam, gel, or cream), bilateral tubal ligation, hysterectomy, bilateral oophorectomy; intrauterine device (IUD) with or without hormones in place or hormonal contraception (oral, injectable, implantable, transdermal, or vaginal) used consecutively for at least 3 months prior to the Screening visit; vasectomized partner or bilateral insertion of Essure® implants for at least 6 months prior to the Screening visit; or postmenopausal status with amenorrhea (no menses) for at least 1 year prior to the Screening visit.
2. Subjects must be willing to refrain from consuming the spice turmeric or any dietary supplements containing turmeric or curcumin (except for the study products) throughout the entire study.
3. Subjects must be available for and willing to attend all evaluation visits.
4. Subjects must be able and willing to give informed consent.
5. Subjects participating in prior studies evaluating CurQ+® or curcumin can participate in the present study so long as they are not currently taking a curcumin containing supplement (including turmeric) and have not done so for 14 days prior to screening.

Exclusion Criteria:

1. Subject is currently receiving therapy with remission-inducing drugs (i.e. methotrexate, TNF biologics, etc.), immunosuppressive drugs (i.e. corticosteroids, transplantation medications, etc.).
2. Subjects must not have taken turmeric- or curcumin-containing dietary supplements within 14 days prior to screening evaluation.
3. Subject has been diagnosed with any clinically significant confounding metabolic disease or condition that would interfere with the study evaluation, as judged by the clinical investigator (slow or fast metabolism resulting from hypo- or hyper-thyroidism, Cushing's Syndrome, Diabetes (except for fully resolved gestational diabetes), etc.) or any conditions that would affect absorption in the GI tract (i.e. inflammatory bowel disease, celiac disease, Behçet's Syndrome, systemic sclerosis, etc.).
4. Subject has known allergy to any of the investigational products, including but not limited to turmeric, curcumin, coconut or coconut oil. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study.
5. Subject's body weight is greater than 300 pounds (136.1 kg) at the time of Screening.
6. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of the first baseline evaluation.
7. Pregnant and/or breastfeeding women, or women who intend to become pregnant during the course of the study.
8. Subject has a history or positive test result of HIV, hepatitis B or hepatitis C.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Comparative effect of differing serum sample preparation methodologies on curcumin absorption levels | 6 hours
  direct analysis versus enzymatic hydrolysis pre-treatment of serum samples to determine Area Under the Curve (AUC) levels in ng-hr/mL of curcumin glucuronide, curcumin sulfate, and free curcumin

SECONDARY OUTCOMES:
Enhanced absorption of BIOCURC compared to standard 95% curcumin powder | 6 hours
  direct analysis of experimental treatment versus active comparator serum samples to determine Area Under the Curve (AUC) levels in ng-hr/mL curcumin glucuronide, curcumin sulfate, and free curcumin

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J. Ruff, Ph.D., Study Director — Stratum Nutrition
Locations (1):
- QPS Bio-Kinetic, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stohs SJ, Chen CYO, Preuss HG, Ray SD, Bucci LR, Ji J, Ruff KJ. The fallacy of enzymatic hydrolysis for the determination of bioactive curcumin in plasma samples as an indication of bioavailability: a comparative study. BMC Complement Altern Med. 2019 Nov 4;19(1):293. doi: 10.1186/s12906-019-2699-x. PMID 31684927
- See also: Evaluation of Increased Absorption of a Curcumin Emulsion (BIOCURC) in Healthy Volunteers — https://bmccomplementalternmed.biomedcentral.com/articles/10.1186/s12906-019-2699-x